CLINICAL TRIAL: NCT00162565
Title: Beta-Blocker Continuation Versus Interruption in Patients With Congestive Heart Failure Hospitalized for Heart Failure Worsening (B-CONVINCED)
Brief Title: Beta-Blocker Continuation Versus Interruption in Heart Failure Worsening
Acronym: BConvinced
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Isabelle. BRINDEL, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P030414
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2009-05-25 (Estimated); Status verified 2005-08

CONDITIONS: Heart Failure, Congestive
Keywords: Heart Failure, Congestive; beta-Adrenergic Blockers
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): bbloquant treatment
  Interventions: Drug: beta-blocker treatment

INTERVENTIONS:
Drug: beta-blocker treatment — beta-blocker treatment

SUMMARY:
The objective of the B-Convinced study is to demonstrate the non-inferiority of beta-blocker continuation compared to its interruption in patients with congestive heart failure who are treated by a beta-blocker and present with an episode of heart failure worsening with pulmonary oedema requiring hospital admission.

162 patients will be randomized in cardiology centers in France. Clinical status (primary endpoint) will be evaluated with a standardized questionnaire 3 days after hospital admission.

DETAILED DESCRIPTION:
Therapeutic strategy of beta-blocker treatment during an episode of heart failure worsening remains unclear. The objective of the B-Convinced study is to demonstrate that continuation of beta-blocker treatment in case of hospitalisation for heart failure worsening is as safe as the interruption of such treatment.

Hypothesis: The proportion of patients clinically improving within 3 days is not inferior when beta-blocker treatment is maintained compared to beta-blocker interruption in case of hospitalisation for heart failure worsening with pulmonary oedema.

Design: Open, randomized non-inferiority trial on two parallel groups of patients. Randomization performed centrally with a vocal server.

Tested Hypothesis: 90% of success in the interruption group, power of 80%, non-inferiority limit of 15% (relative reduction). 162 patients are required with such a hypothesis.

Primary Endpoint: Clinical improvement within 3 days of hospital admission evaluated by the investigator by a standardized questionnaire.

Secondary Endpoints: Clinical improvement at day 8 or at hospital discharge, morbidity-mortality at 4 months.

34 participating centres in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure treated with beta-blocker; hospitalisation for heart failure worsening with pulmonary oedema.
* Left ventricular ejection fraction less than 40%

Exclusion Criteria:

* Indication of intravenous positive inotropic treatment
* Indication to withdraw beta-blocker treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2004-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Clinical status (questionnaire): the percentage (%) of patients with clinical improvement is the primary endpoint criterion. | at day 3 of hospital admission

SECONDARY OUTCOMES:
Clinical status (evaluation by investigator and autoevaluation by patient) | at day 8 after hospital admission
BNP change | between admission, day 3 and day 8
Mortality, hospital admission, % of patients with beta-blocker treatment | at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe P Lechat, MD, PhD, Study Director — Hopital Pitie-Salpetriere, Paris, France; Guillaume Jondeau, MD, PhD, Principal Investigator — Hopital Ambroise-Pare, Boulogne, France
Locations (32):
- France (32):
  - Hôpital Victor Dupuy, Argenteuil
  - Les Etablissements Hospitaliers du Bessin, Bayeux
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Centre Hospitalier Universitaire de Caen, Caen
  - Hôpital Fontenoy de Chartres, Chartres
  - Centre Hospitalier de Cholet, Cholet
  - Hôpital Antoine Béclère, Clamart
  - Hôpital Beaujon, Clichy
  - Hôpital de Corbeil, Corbeil
  - Hôpital Henri Mondor, Créteil
  - Hôpital du Bocage, Dijon
  - Hôpital A. Michallon, Grenoble
  - Centre Hospitalier de Versailles, Le Chesnay
  - Hôpital Saint-Philibert, Lomme
  - Hôpital Saint-Joseph Saint-Luc, Lyon
  - Hôpital de la Timone, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpital René Laënnec, Nantes
  - Hôpital Pasteur, Nice
  - Hôpital des Armées du Val de Grâce, Paris
  - Hôpital Lariboisière, Paris
  - Groupe Hospitalier Pitié-Salpêtrière, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Saint-Michel, Paris
  - Centre Hospitalier Universitaire La Milétrie, Poitiers
  - Centre Hospitalier Regional Dubos, Pontoise
  - Centre Hospitalier Universitaire Potcaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Centre Hospitalier Universitaire Hautepierre, Strasbourg
  - Hôpital de Rangueil, Toulouse
  - Hôpital Trousseau, Tours
  - Hôpital de Brabois, Vandœuvre-lès-Nancy